CLINICAL TRIAL: NCT00864045
Title: A Randomised, Double-blind, Parallel-group, Flexible-dose Trial Evaluating the Efficacy and Safety of 12 Weeks of Treatment With Sertindole or Olanzapine in Patients With Schizophrenia in Asia
Brief Title: Sertindole in Asian Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11286
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — sertindole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertindole (Experimental)
  Interventions: Drug: Sertindole
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Sertindole — Sertindole flexible doses per os, 12, 16 or 20mg/day according to response and tolerability, initially up-titrated from 4mg/day to target dose 16mg/day within the first 16 days
  Arms: Sertindole
Drug: Olanzapine — Olanzapine flexible doses per os, 10, 15 or 20mg/day according to response and tolerability, initially up-titrated from 10mg/day to target dose 15mg/day within the first 16 days
  Arms: Olanzapine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of sertindole in patients with schizophrenia in Asia.

DETAILED DESCRIPTION:
This study is the first randomised clinical trial performed in Asia with sertindole, aiming at comparing sertindole efficacy and safety to that of another atypical antipsychotic.

Sertindole is a limbic-selective antipsychotic agent with a unique neuropharmacological profile. Sertindole has shown significant improvements relative to placebo against both positive and negative symptoms of schizophrenia (measured by PANSS total, PANSS negative and positive subscale scores). It is well tolerated and shows placebo-level incidence of extrapyramidal symptoms (EPS). Sertindole is associated with a dose-dependent increase in the QT interval, but this does not translate into an excess mortality with sertindole relative to that of other recently developed antipsychotics in their respective clinical development programmes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18-65 years (extremes included), suffering from schizophrenia
* Positive and Negative Syndrome Scales (PANSS) total score between 60 and 120 (extremes included) at screening and baseline
* Based on the patient's clinical status, an antipsychotic treatment is indicated
* Otherwise healthy
* Female patients of non-childbearing potential, or non-pregnant, not breast-feeding women of childbearing potential, using adequate birth control methods

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than schizophrenia
* Has never before received antipsychotic drugs
* Has received a depot antipsychotic medication within less than one dose interval prior to Screening
* History of clinically significant cardiovascular disease, congestive heart failure, cardiac hypertrophy, arrhythmia or bradycardia (<50 beats per minute)
* Congenital long QT syndrome or a family history of this disease, or in patients with known acquired QT interval prolongation (QTc above 450 msec in males and 470 msec in females at Screening)
* Significant risk of suicide and/or violent behaviour
* Known history of narrow angle glaucoma
* Substance or alcohol abuse, current alcohol dependence
* Use of disallowed concomitant medication

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of 12 weeks treatment with flexible doses of sertindole in comparison to flexible doses of olanzapine in patients with schizophrenia. | 12 weeks

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of 12 weeks treatment with flexible doses of sertindole in comparison to flexible doses of olanzapine in patients with schizophrenia. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CN001, Beijing, China

REFERENCES:
- [Derived] Kim EY, Chang SM, Shim JC, Joo EJ, Kim JJ, Kim YS, Ahn YM. Long-term effectiveness of flexibly dosed paliperidone extended-release: comparison among patients with schizophrenia switching from risperidone and other antipsychotic agents. Curr Med Res Opin. 2013 Oct;29(10):1231-40. doi: 10.1185/03007995.2013.816277. Epub 2013 Jul 16. PMID 23777311